CLINICAL TRIAL: NCT06531642
Title: Comparison of Early Proton Pump Inhibitor Initiation Versus Usual Care on Acute Kidney Injury (CEPU-AKI) in Hemorrhagic Shock Patients: a Prospective Randomized Controlled Trial
Brief Title: Comparison of Early Proton Pump Inhibitor Initiation Versus Usual Care on Acute Kidney Injury in Hemorrhagic Shock Patients
Acronym: Trauma AKI PPI
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, yafen liang, M.D., Professor, Chief of Division of Cardiovascular Anesthesiology, Vice Chair of Clinical Research, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-24-0411; 175191 (Other Grant/Funding Number: Trauma Research and Combat Casualty Care Collaborative (TRC4))
Record Dates: First submitted 2024-07-19; First posted 2024-08-01 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; AKI; Proton Pump Inhibitors; Hemorrhagic Shock; Trauma Patients; PPI; Randomized Controlled Trial
MeSH Terms: conditions — Acute Kidney Injury; Shock, Hemorrhagic | interventions — Pantoprazole

STUDY DESIGN:
Intervention Model Description: Study group patients will receive pantoprazole early (40 mg iv q12H, within 2 hours of ED arrival and after study enrollment) and control group patients will receive the usual timing (40 mg iv daily, at routine timing, usually in the intensive care unit), then for 2 additional days after the initial injury insult.
Who Masked: Outcomes Assessor
Masking Description: Partial blinded, only the laboratory testing technician/outcome assessor will be blinded to the study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Initiation (Experimental): Within 2 hours of emergency department (ED) admission after inclusion criteria is met, administer 1st dose of Protonix (pantoprazole) 40 mg, then followed by 40 mg q12hrs for 2 additional days
  Interventions: Drug: Protonix (Pantoprazole) 40 mg q 12 hrs for 2 days
- Usual Care (Active Comparator): Administer 1st dose of 40 mg Protonix (pantoprazole) at the usual timing (current practice: in the intensive care unit), then followed by 40 mg daily for 2 additional days.
  Interventions: Drug: Protonix (pantoprazole) 40 mg q 24 hrs for 2 days

INTERVENTIONS:
Drug: Protonix (Pantoprazole) 40 mg q 12 hrs for 2 days — Within 2 hours of ED admission after inclusion criteria is met, administer 1st dose of Protonix (pantoprazole) 40mg, then followed by 40mg q12hrs for 2 additional days.
  Arms: Early Initiation
Drug: Protonix (pantoprazole) 40 mg q 24 hrs for 2 days — Administer 1st dose of 40mg Protonix (pantoprazole) at the usual timing (current practice: in the intensive care unit), then followed by 40mg daily for 2 additional days.
  Arms: Usual Care

SUMMARY:
The investigators propose a single-center, randomized, controlled trial to determine whether early initiation of proton pump inhibitor (PPI), pantoprazole, will decrease acute kidney injury (AKI) for trauma patients presenting with hemorrhagic shock compared to routine timing of initiation of PPI. Kidney injury will be assessed by the urinary kidney injury biomarkers, and the incidence, severity and AKI-free days within first week and major adverse kidney events (MAKE) at day 30. The specific aims of the study will be achieved by a cohort of 100 patients to receive either early(study) or routine (control) administration of pantoprazole for 2 days after the initial injury insult.

DETAILED DESCRIPTION:
Traumatic injuries account for 10% of all deaths globally and are the leading cause of mortality for trauma patients under 46 in the United States. Hemorrhage is the primary cause of death in both civilian and military trauma scenarios worldwide. Following hemorrhage and traumatic brain injury, organ failure, including acute kidney injury (AKI), is the third leading cause of death in trauma patients. AKI occurs in up to 50% of patients with hemorrhagic shock and is linked to increased morbidity, extended hospital stays, progression to chronic kidney disease, and higher short- and long-term mortality rates. Even patients with mild AKI, as classified by the RIFLE criteria (Risk, Injury, Failure, Loss of kidney function, and End-stage kidney disease), face a 2.5 times higher risk of mortality. Battlefield conditions often delay access to definitive medical care for injured soldiers, highlighting the urgent need for effective shock treatments to minimize organ damage, such as AKI.

The investigators propose a single-center, randomized, controlled trial to determine whether early initiation of proton pump inhibitor (PPI), pantoprazole, will decrease acute kidney injury (AKI) for trauma patients presenting with hemorrhagic shock compared to routine timing of initiation of PPI.

Our study will include adults (over 18 years old) who meet the criteria for hemorrhagic shock, as these patients are more susceptible to hypoxic kidney damage due to bleeding and hypovolemia. This will allow us to assess whether early PPI initiation can better protect the kidneys during the early stages of hypoxic damage.

To evaluate this, the investigators will measure urinary kidney injury biomarkers in trauma patients to compare early pantoprazole initiation (study group) with the usual timing of PPI initiation (control group) (n=100, primary endpoint). Additionally, the investigators will assess whether early pantoprazole initiation decreases the incidence, severity, and number of AKI-free days within the first week post-hemorrhagic shock, as well as major adverse kidney events (MAKE: a composite of death, dialysis, renal hospitalization, or sustained kidney dysfunction) 30 days after the initial injury.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years of age)
* Patient meets hemorrhagic shock criteria:
* Hypovolemic shock from traumatic acute bleeding
* Systolic blood pressure ≤ 90 mmHg AND tachycardia (HR ≥ 108) at presentation to the ED; OR
* Systolic blood pressure ≤ 70 mmHg at presentation to the ED.

Exclusion Criteria:

* Patients <18 years of age
* Patients known to be actively on renal replacement therapy
* Cardiac arrest prior to ED arrival or who are deemed to have expected survival of less than 24 hours
* History of PPI sensitivity or allergy
* Patient who are already enrolled in other trials prior to ED arrival and these trials do not allow co-enrollment
* Patient who presents with ongoing GI bleeding that will require higher dose of GI prophylaxis
* Vulnerable populations such as pregnant women and prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-07 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Urinary Kidney Biomarker Levels | From enrollment until 48 hours after injury
  The investigators will measure the urinary kidney biomarker KIM-1 (kidney injury molecule-1) levels at the different time points of urine sample collection (baseline, 8 hrs, 24 hrs and 48 hrs)

SECONDARY OUTCOMES:
Acute Kidney Injury Staging | From enrollment until 5 days of initial injury
  The investigators will classify each patient to an AKI stage (1, 2 or 3) according to the 2012 Kidney Disease Improving Global Outcomes (KDIGO) which uses creatinine levels and estimated glomerular filtration rate (eGFR) levels each day for 5 days after enrollment.
Major Adverse Kidney Events | From enrollment until 30 days of initial injury
  The investigators will follow up on patients enrolled in the study and ask about patient demise, necessity of dialysis of any type, hospitalizations due to renal problems, or sustained kidney dysfunction after 30 days of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Yafen Liang, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Texas Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No